CLINICAL TRIAL: NCT01057875
Title: The Effects of Caffeine on Exhaled Nitric Oxide Levels and Methacholine PC20
Brief Title: Effects of Caffeine on Methacholine Challenge and Exhaled Nitric Oxide Levels.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Donald Cockcroft, MD, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BIO REB 09-186
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2010-10-07 (Estimated); Status verified 2010-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- coffee with caffeine (Experimental)
  Interventions: Other: caffeine
- decaffeinated coffee (Placebo Comparator): Starbuck's Grande Pike Roast Decaf
  Interventions: Other: No caffeine

INTERVENTIONS:
Other: caffeine — Starbuck's Grande Pike Roast coffee
  Arms: coffee with caffeine
Other: No caffeine — Starbuck's Grande Pike Roast Decaffeinated Coffee
  Arms: decaffeinated coffee

SUMMARY:
To investigate whether or not the ingestion of caffeine with alter airway responsiveness to methacholine and/or change the level of exhaled nitric oxide.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of asthma
* FEV1 greater than 65%

Exclusion Criteria:

* asthma is poorly controlled
* presence of other airway disease (e.g. COPD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
methacholine pc20 | 1 hour post ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Donald W Cockcroft, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Derived] Yurach MT, Davis BE, Cockcroft DW. The effect of caffeinated coffee on airway response to methacholine and exhaled nitric oxide. Respir Med. 2011 Nov;105(11):1606-10. doi: 10.1016/j.rmed.2011.06.006. Epub 2011 Jul 2. PMID 21726992